CLINICAL TRIAL: NCT07334366
Title: A 12-week Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Broccoli Sprout Extract on Cognitive Function Improvement in Adults With Mild Cognitive Impairment
Brief Title: Broccoli Sprout Extract for Cognitive Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12-2024-018
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Dysfunction; Cognitive Decline
Keywords: cognition
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broccoli group (Experimental): This group takes broccoli sporout extract for 12 weeks.
  Interventions: Dietary Supplement: Broccoli sprout extract (BSE)
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo Control

INTERVENTIONS:
Dietary Supplement: Broccoli sprout extract (BSE) — BSE 1,000 mg/day for 12 weeks
  Arms: Broccoli group
Dietary Supplement: Placebo Control — Placebo (crystalline cellulosel) 1,000 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
This clinical trial aims to determine whether broccoli sprout extract improves cognitive function in adults with mild cognitive impairment and to assess its safety.

The main questions are:

* Does broccoli sprout extract improve cognitive function in participants?
* What side effects occur when participants take broccoli sprout extract?

DETAILED DESCRIPTION:
Researchers will compare broccoli sprout extract to a placebo to evaluate their effectiveness in improving cognitive function in participants.

Participants will:

* Take dietary broccoli sprout extract or a placebo daily for 12 weeks.
* Visit the clinic at screenig, 0, 6, and 12 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults aged 55-85 years (inclusive), both male and female
* Global Deterioration Scale (GDS) score of 2-3:

GDS 2: Subjective memory impairment without objective evidence GDS 3: Mild objective memory impairment

* Absence of dementia according to established diagnostic criteria
* Ability to read Korean

Exclusion Criteria:

* Severe medical conditions within the past 6 months: History of severe cerebrovascular disease (cerebral infarction, cerebral hemorrhage), cardiac disease (angina, myocardial infarction, heart failure, arrhythmia requiring treatment), or malignancy (Note: Participants with a history of cerebrovascular or cardiac disease who are clinically stable may be included at the investigator's discretion)
* Cognitive impairment-associated diseases: Dementia, Parkinson's disease, cerebral infarction, or other conditions associated with cognitive decline Uncontrolled hypertension: Blood pressure ≥160/100 mmHg (measured after 10 minutes of rest)
* Poor glycemic control: Fasting blood glucose ≥160 mg/dL in diabetic patients
* Uncontrolled thyroid dysfunction: Currently receiving treatment for uncontrolled hypothyroidism or hyperthyroidism
* Renal impairment: Serum creatinine ≥2 times the upper limit of normal for the institution
* Hepatic impairment: AST or ALT ≥2 times the upper limit of normal for the institution
* Severe gastrointestinal symptoms: Complaints of severe heartburn, dyspepsia, or other gastrointestinal distress
* Medications affecting cognitive function within the past month: Use of drugs (antipsychotics, anti-degenerative agents, cognitive enhancers, tricyclic antidepressants, hormone replacement therapy) or health functional foods that may influence cognitive function due to dementia or other cognitive abnormalities
* Other clinical trial participation: Participation in other drug clinical trials within the past month or planned participation during the study period
* Alcohol use disorder, severe
* Food allergies: Known allergic reactions to study product components
* Investigator discretion: Any other condition deemed inappropriate for study participation by the investigator

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 12 weeks in total Computerized NeuroCognitive Function Test score comprising verbal learning test, digit span test, and auditory continuous performance test | 12 weeks
  The change in total CNT score from baseline to 12 weeks, calculated as the sum of verbal learning test, digit span test, and auditory continuous performance test scores. Higher total CNT scores indicate better neurocognitive function across the domains of memory, attention, and sustained concentration. This composite measure assesses overall cognitive performance, where positive changes (increase in total score) indicate cognitive improvement and negative changes (decrease in total score) suggest cognitive decline.

SECONDARY OUTCOMES:
Change from baseline to 12 weeks in verbal learning test score | 12 weeks
  The change in verbal learning test score from baseline to 12 weeks, measuring memory and learning capacity. Higher scores indicate better verbal memory and learning ability. This assessment evaluates the ability to acquire, retain, and recall verbal information over multiple learning trials. Positive changes (increase in score) indicate improvement** in verbal memory function, while negative changes (decrease in score) suggest a decline in verbal learning capacity.
Change from baseline to 12 weeks in digit span test score | 12 weeks
  The change in digit span test score from baseline to 12 weeks, measuring working memory and attention span. Higher scores indicate better working memory and attention capacity. This assessment evaluates the ability to temporarily hold and manipulate numerical information in memory through forward and backward digit recall tasks. Positive changes (increase in score) indicate improvement in working memory capacity, while negative changes (decrease in score) suggest decline in attention and short-term memory function.
Change from baseline to 12 weeks in auditory continuous performance test score | 12 weeks
  The change in auditory continuous performance test score from baseline to 12 weeks, measuring sustained attention and concentration abilities. Higher scores indicate better sustained attention and concentration capacity. This assessment evaluates the capacity to maintain focused attention and respond appropriately to auditory stimuli over an extended period. Positive changes (increase in score) indicate improvement in sustained attention function, while negative changes (decrease in score) suggest decline in concentration and vigilance capabilities.
Change from baseline to 12 weeks in Korean Mini-Mental State Examination (MMSE-K) total score | 12 weeks
  The change in MMSE-K total score from baseline to 12 weeks, providing a brief assessment of global cognitive function. Higher scores indicate better global cognitive function. This standardized instrument evaluates orientation, attention, memory, language, and visuospatial abilities. Positive changes (increase in score) indicate improvement in overall cognitive status, while negative changes (decrease in score) suggest decline in cognitive function.
Change from baseline to 12 weeks in serum brain-derived neurotrophic factor (BDNF) concentration | 12 weeks
  The change in serum BDNF concentration from baseline to 12 weeks, measured in ng/mL or pg/mL. BDNF is a neurotrophin that plays a crucial role in neuronal survival, growth, and synaptic plasticity. Positive changes indicate increased BDNF levels associated with enhanced neuroplasticity and neuroprotection, while negative changes suggest decreased neurotrophic support.
Change from baseline to 12 weeks in serum malondialdehyde (MDA) concentration | 12 weeks
  The change in serum MDA concentration from baseline to 12 weeks, measured in μmol/L or nmol/mL. MDA is a biomarker of lipid peroxidation and oxidative stress, reflecting cellular damage from reactive oxygen species. Positive changes indicate increased oxidative stress and cellular damage, while negative changes stress and improved antioxidant status.
Change from baseline to 12 weeks in serum superoxide dismutase (SOD) activity | 12 weeks
  The change in serum SOD activity from baseline to 12 weeks, measured in U/mL or U/mg protein. SOD is a key antioxidant enzyme that catalyzes the dismutation of superoxide radicals, providing cellular protection against oxidative damage. Positive changes indicate enhanced antioxidant capacity and cellular protection, while negative changes suggest reduced antioxidant defense mechanisms.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea